CLINICAL TRIAL: NCT00002940
Title: Hydroxyurea Treatment of EBV-Associated Primary CNS Lymphoma in Children and Adults With AIDS
Brief Title: Hydroxyurea in Treating Patients With Epstein-Barr Virus-Associated Primary CNS Lymphoma and AIDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065389; SJCRH-DID-965 (Other: St. Jude Children's Research Hospital); NCI-V97-1143 (Other: National Cancer Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-11-24 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2002-06

CONDITIONS: Lymphoma
Keywords: AIDS-related primary CNS lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: hydroxyurea

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of hydroxyurea in treating patients with Epstein-Barr virus-associated primary CNS lymphoma and AIDS.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the objective response rate of PCNSL in AIDS patients treated with hydroxyurea. II. Investigate whether levels of Epstein-Barr virus (EBV) DNA in the blood or cerebral spinal fluid are correlates of PCNSL disease activity.

OUTLINE: This is an open label pilot study. Patients receive oral hydroxyurea tid. A course of hydroxyurea consists of 4 weeks of therapy. On day 28, after the first course of treatment, tumor size is analyzed by MRI. If no reduction in tumor size is seen on day 28, hydroxyurea dose is increased. If a CR or PR is demonstrated, patients continue on the same treatment at the original dose. MRI evaluation is again taken on day 56 of treatment. Patients with progressive disease at this evaluation are considered to have no treatment response.

PROJECTED ACCRUAL: 15-25 patients will be enrolled. Approximately 8-10 patients will be accrued annually.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven EBV-associated primary CNS lymphoma HIV infection confirmed by a positive ELISA and Western blot

PATIENT CHARACTERISTICS: Age: Open to children and adults of any age Performance Status: Karnofsky at least 50% Life Expectancy: At least 4 weeks Hematopoietic: Hemoglobin at least 6.9 gm/dL ANC at least 500/mm3 Platelet count at least 50,000/mm3 Hepatic: Bilirubin no greater than 1.5 x upper limit of normal (ULN) (1.5 to 2.5 x ULN if receiving indinavir) Renal: Creatinine no greater than 1.5 x ULN Cardiovascular: Not specified Other: Not pregnant or nursing Contraception required in fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: Prior or concurrent antiretroviral therapy allowed No prior EBV-associated primary CNS lymphoma therapy within 1 week of study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-10; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen S. Slobod, MD, Study Chair — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Saint Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org